CLINICAL TRIAL: NCT00999674
Title: The Effect of an Exercise Program on the Health-quality of Life (HQL) in Older
Brief Title: The Effect of an Exercise Program on the Health-quality of Life (HQL) in Older Adults
Acronym: HQL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahrekord University (Other)
Responsible Party: Health Ministry, Faculty of Medicine
Allocation: Randomized | Purpose: Health Services Research
Other Study IDs: 4113
Record Dates: First submitted 2009-10-18; First posted 2009-10-22 (Estimated); Last update posted 2009-10-22 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
Keywords: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: An exercise program — The study subjects were recruited among those who responded to advertisements in outpatient clinics

SUMMARY:
The present study aimed to investigate the effect of exercise program on health-quality of life (HQL) in older adults.

DETAILED DESCRIPTION:
The questionnaire consisted of demographic data (such as age, gender, educational level, and employment) and the LEIPAD questionnaire used to measure HQL.

ELIGIBILITY:
Inclusion Criteria:

* sixty healthy adults volunteers
* over the age of 55 years

Exclusion Criteria:

* neurological disorder
* acute heart impairment
* unstable chronic illness
* severe musculo-skeletal impairment

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Saeed Heydarnejad, PhD, Principal Investigator — Health Ministry

REFERENCES:
- [Derived] Heydarnejad S, Dehkordi AH. The effect of an exercise program on the health-quality of life in older adults. A randomized controlled trial. Dan Med Bull. 2010 Jan;57(1):A4113. PMID 20175947